CLINICAL TRIAL: NCT03186599
Title: Analysis of Initial Adherence and Its Impact on Long-term Adherence to Hormonal Therapy for Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gachon University (Other)
Collaborators: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yul Ha Min, Assistant professor, Gachon University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-0351
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
Keywords: Medication Event Monitoring System; adherence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high adherence control group (No Intervention): -Patients on continuous MEMS monitoring with usual care.
- low adherence control group (No Intervention): -Patients on continuous MEMS monitoring with usual care.
- low adherence intervention group (Experimental): * Patient with the WALKON mobile application.
  * Patient with monthly feedback call
  * Patients on continuous MEMS monitoring.
  Interventions: Behavioral: low adherence intervention group

INTERVENTIONS:
Behavioral: low adherence intervention group — Monthly, the study coordinator will give calls to encourage physical activities and medication adherence using MEMS and WALKON activity data.
  Arms: low adherence intervention group

SUMMARY:
A trial will be conducted on 200 breast cancer patients with adjuvant hormonal therapy. The study included 6 months baseline measurement, and 12 months intervention. Patients will be assigned to high adherence or low adherence group. Then, through randomization, low adherence patients will be assigned to the intervention or control group. Study Coordinator delivers the intervention using the WALKON mobile application. Control participants receive usual care with continuous monitoring using Medication Event Monitoring System (MEMS) device.

DETAILED DESCRIPTION:
* Baseline measurement (n=200): screening and enrollment
* 3-month visit: collecting MEMS data
* 6-month visit: collecting MEMS data and assigned to the high adherence (n=70) or low adherence group (n=75). The low adherence intervention group (n=75) will be educated about the WALKON mobile application.
* 12-month visit: Control group: collecting MEMS data intervention group: monthly calls + collecting MEMS data
* 18-month visit: collecting MEMS data and interview

ELIGIBILITY:
Inclusion Criteria:

* Stage 0-III breast cancer
* Treated with Adjuvant hormonal therapy

Exclusion Criteria:

* Stage IV breast cancer
* Breast cancer recurrence or metastasis
* Severe medical illness

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-06-08 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
physical activity (daily steps) | 12 months
  Comparison of daily steps using WALKON application

SECONDARY OUTCOMES:
Medication adherence using MEMS device | 18 months
  Comparison of adjuvant hormonal therapy adherence using MEMS device

CONTACTS AND LOCATIONS:
Overall Officials: Yul ha Min, PhD, Principal Investigator — Gachon University
Locations (1):
- Asan Medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided